CLINICAL TRIAL: NCT05108532
Title: Polish Revision Obesity Surgery Study
Acronym: PROSS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical University of Gdansk (Other)
Collaborators: University of Warmia and Mazury in Olsztyn (Other); Jagiellonian University (Other); Medical University in Białystok (Unknown); Nicolaus Copernicus University (Other); Military Institute od Medicine National Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PROSS
Record Dates: First submitted 2021-10-25; First posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Metabolic Disease; Obesity, Morbid
Keywords: bariatric surgery failure; revisional bariatric surgery; secondary bariatric procedure
MeSH Terms: conditions — Metabolic Diseases; Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients after revisional bariatric surgery.: This cohort will include patients, who underwent revisional bariatric surgery.

SUMMARY:
Bariatric surgery is well established method of treating patients with obesity. Obesity is well-documented risk factor for many health conditions including some cancer, cardiovascular diseases, pulmonary diseases and type-2 diabetes. Bariatric surgery is associated with improved comorbidities, quality of life and survival in severe obesity. However, the rate of conversion or revisional bariatric surgeries is increasing nowadays. Recent date estimate the rate of revisional procedures between 8-25% of all bariatric surgeries performed worldwide.

Weight recidivism or fail to achieve a significant weight loss (estimated 10-20% of operated patients) remains a challenge for surgeons and patients. This has economic and health implications, leading to reduction in quality of life and increased prevalence of obesity-related comorbid conditions. Therefore, the aim of this study is to identified patients with failure after primary bariatric procedure in population of Poland.

DETAILED DESCRIPTION:
All participating medical institutions performing metabolic and bariatric surgeries from Poland can register patients via online questionaries. The database will include all patients with full preoperative history regarding the status of comorbidities, maximum weight and BMI. Details regarding initial surgery will be collected: type of procedure, time of procedure, length of the procedure, technical aspects (type of anastomosis, location of the anastomosis, type and amount of staplers used, length of bypassed jejunum, type of gastric band), length of hospital stay, short-term complications. The outcomes of initial surgery will be noticed: %TWL, minimum weight and BMI, remission of comorbidities, improvement of comorbidities, reduction of pharmacological treatment. Long-term postoperative complications in example de novo reflux, stenosis of anastomosis, stricture of gastric pouch will be included in analysis. The cause of revisionary surgery will be analyzed. The secondary bariatric procedure will be analyzed in terms of time, type and its length. Detail information of technical aspects will be collected. The complications and outcomes of revisional surgery will be acquired from hospitals registers, as well as, informations received from clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

Patients after revisional bariatric surgery, male and females over 18 years old, any type of primary bariatric surgery.

Exclusion Criteria:

Lack of follow-up, lack of anthropometric details at any point of a study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after revisionary bariatric and metabolic surgery. Operated in Poland.m
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
indications for revisional bariatric operations, | 10 years
type of surgeries most frequently chosen as revisional procedures | 10 years
course of perioperative treatment among patients undergoing revisional and secondary revisional bariatric surgery | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Monika Proczko-Stepaniak, Prof, Principal Investigator — Medical University of Gdansk
Locations (1):
- Medical University of Gdańsk, Gdansk, Poland

REFERENCES:
- [Background] Switzer NJ, Karmali S, Gill RS, Sherman V. Revisional Bariatric Surgery. Surg Clin North Am. 2016 Aug;96(4):827-42. doi: 10.1016/j.suc.2016.03.004. PMID 27473804
- [Background] Acevedo E, Mazzei M, Zhao H, Lu X, Edwards MA. Outcomes in conventional laparoscopic versus robotic-assisted revisional bariatric surgery: a retrospective, case-controlled study of the MBSAQIP database. Surg Endosc. 2020 Apr;34(4):1573-1584. doi: 10.1007/s00464-019-06917-5. Epub 2019 Jun 17. PMID 31209611
- [Background] van Rijswijk AS, van Olst N, Schats W, van der Peet DL, van de Laar AW. What Is Weight Loss After Bariatric Surgery Expressed in Percentage Total Weight Loss (%TWL)? A Systematic Review. Obes Surg. 2021 Aug;31(8):3833-3847. doi: 10.1007/s11695-021-05394-x. Epub 2021 May 17. PMID 34002289
- [Derived] Dowgiallo-Gornowicz N, Janik M, Lech P, Kowalski G, Major P; PROSS -Collaborative Study Group. Revisional bariatric surgery after adjustable gastric band: a multicenter Polish Revision Obesity Surgery Study (PROSS). BMC Surg. 2023 Apr 20;23(1):94. doi: 10.1186/s12893-023-02002-w. PMID 37081459
- [Derived] Labul M, Wysocki M, Bartosiak K, Orlowski M, Katkowski B, Jaworski P, Malczak P, Major P; PROSS-Collaborative Study Group. Analysis of the Factors Contributing to Bariatric Success After Laparoscopic Redo Bariatric Procedures: Results from Multicenter Polish Revision Obesity Surgery Study (PROSS). Obes Surg. 2022 Dec;32(12):3879-3890. doi: 10.1007/s11695-022-06306-3. Epub 2022 Oct 15. PMID 36242680